CLINICAL TRIAL: NCT04434599
Title: Fluoroscopic, Contact Force and Local Impedance With Ultra-high Density Mapping Guided Radiofrequency Ablation Comparison for cavoTricuspid Isthmus dependenT Atrial fluttER: the FLUTTER Study
Acronym: FLUTTER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Karan Saraf, Investigator, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 281105
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Typical Atrial Flutter
Keywords: radiofrequency ablation; contact force; local impedance

STUDY DESIGN:
Intervention Model Description: 114 patients randomised 1:1:1 to either fluoroscopically guided OR contact force guided OR local impedance guided radiofrequency catheter ablation of typical atrial flutter
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fluoroscopically guided ablation (Active Comparator): These patients will receive one catheter ablation of typical atrial flutter by fluoroscopically guided radiofrequency ablation catheters
  Interventions: Device: Fluoroscopically guided ablation
- Contact force guided ablation (Active Comparator): These patients will receive one catheter ablation of typical atrial flutter by contact force guided radiofrequency ablation catheters using the CARTO 3D electroanatomic mapping system
  Interventions: Device: Contact force guided ablation
- Local impedance guided ablation (Active Comparator): These patients will receive one catheter ablation of typical atrial flutter by local impedence guided radiofrequency ablation catheters using the Rhythmia Ultra-high density 3D electroanatomic mapping system
  Interventions: Device: Local impedance guide ablation

INTERVENTIONS:
Device: Fluoroscopically guided ablation — Catheter ablation of the cavotricuspid isthmus using ablation catheters guided by fluoroscopy
  Arms: Fluoroscopically guided ablation
Device: Contact force guided ablation — Catheter ablation of the cavotricuspid isthmus using ablation catheters guided by contact force measurement and 3D electroanatomic mapping
  Arms: Contact force guided ablation
Device: Local impedance guide ablation — Catheter ablation of the cavotricuspid isthmus using ablation catheters guided by local impedance measurement and ultra-high density 3D electroanatomic mapping
  Arms: Local impedance guided ablation

SUMMARY:
Catheter ablation is a first-line treatment for patients with cavotricuspid isthmus (CTI) dependent atrial flutter (AFL; also known as typical AFL), a common arrhythmia. This is done using radiofrequency (RF) catheters and single-procedure success is approximately 95%. Ablation is often done using one of three methods:

1. fluoroscopically, using X-rays to guide the operator to visualise catheter position within the heart. This method involves the most radiation exposure to patient and operator. Ablation is generally performed for a set time-period (eg. 30-60secs) to ensure each ablation lesion is successful.
2. using a 3-dimensional mapping system which allows the catheters to be magnetically located and visualised on a monitor without X-rays, and using "contact force" (CF) sensing catheters. This requires minimal X-ray use, and by ensuring a minimum degree of force between catheter tip and the heart before applying RF for a set time-period (eg. 30 seconds), operators can be more confident of successful lesions.
3. using an ultra-high density mapping system which uses magnetic tracking as above, but allows higher resolution visualisation of the cardiac electrical system with potential for improving procedure success; this has not yet been formally evaluated for AFL. Catheters using this method use "local impedance" (LI) instead of CF. This is a direct measure of heart tissue impedance with real-time changes during ablation. A minimum drop or plateau in the LI value during ablation allows confidence of lesion success, without the need to ablate for a pre-defined time-period. This could potentially reduce ablation time and subsequent complications, but has also not yet been formally compared to the above for this indication.

This prospective randomised study aims to compare these three standard of care procedures to determine if differences in ablation metrics, efficacy and safety exist.

ELIGIBILITY:
Inclusion Criteria:

* Patients under the care of the NHS
* Aged 18-80 years
* Symptoms and 12-lead ECG suggestive of typical (cavotricuspid isthmus dependent) atrial flutter
* Due to undergo first-time cavotricuspid isthmus ablation (including as part of a combined ablation if also having pulmonary vein isolation for atrial fibrillation) on clinical grounds

Exclusion Criteria:

Pre-procedure:

* Inability to given informed consent / lack of mental capacity
* Obesity (BMI >40)
* Congenital heart disease or tricuspid valve abnormalities likely to prolong procedure time, including Ebstein anomaly, atrial septal defects, tricuspid valve repair or replacement, severe tricuspid valve regurgitation
* Inability or unwillingness to receive oral anticoagulation with a vitamin K antagonist (VKA) or non-VKA oral anticoagulant (NOAC)
* Previous cavotricuspid isthmus ablation procedure
* Known infiltrative cardiomyopathy
* Pregnancy
* Age < 18 or >80
* Inability to speak adequate English/need for an interpreter for study consent process

Post procedure:

- arrhythmia mechanism found not to be cavotricuspid isthmus dependent atrial flutter

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-30 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Time from first application of radiofrequency energy to confirmation of bidirectional cavotricuspid isthmus block | At time of procedure
  Time from first application of radiofrequency energy to confirmation of bidirectional cavotricuspid isthmus block

SECONDARY OUTCOMES:
Mean total ablation time to achieve bidirectional cavotricuspid isthmus block | At time of procedure
  Mean total ablation time to achieve bidirectional cavotricuspid isthmus block
Mean total radiation exposure | At time of procedure
  Mean total radiation exposure
Mean total number of ablation lesions required to achieve bidirectional cavotricuspid isthmus block | At time of procedure
  Mean total number of ablation lesions required to achieve bidirectional cavotricuspid isthmus block
Number of cases where bidirectional cavotricuspid isthmus block was not achieved after the first pass of ablation | At time of procedure
  Number of cases where bidirectional cavotricuspid isthmus block was not achieved after the first pass of ablation
Mean time taken for second pass ablation (with or without the use of 3D mapping) to achieve bidirectional cavotricuspid isthmus block | At time of procedure
  Mean time taken for second pass ablation (with or without the use of 3D mapping) to achieve bidirectional cavotricuspid isthmus block
Locations of breakthrough across the initial ablation line | At time of procedure
  Locations of breakthrough across the initial ablation line
Frequency of procedural complications | At time of and immediately following procedure
  Frequency of procedural complications
Acute and medium-term success rates | 12 months
  Acute and medium-term success rates

IPD SHARING:
Plan to Share IPD: No